CLINICAL TRIAL: NCT01308827
Title: Continuation of the Costa Rican Epidemiologic Surveillance for Invasive Pneumococcal Disease After Introduction of the Seven Valent Vaccine Into the Universal Vaccination Program
Brief Title: Costa Rica Epidemiological Study on S. Pneumoniae
Status: Suspended | Type: Observational
Why Stopped: Study recruitment was suspended due to lack of funding
Sponsor: Instituto de Atención Pediátrica (Other)
Collaborators: Ben-Gurion University of the Negev (Other); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: IAP-036; IAP-036 (Other: Instituto de Atencion Pediatrica)
Record Dates: First submitted 2011-02-25; First posted 2011-03-04 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Streptococcus Pneumoniae
Keywords: Children 28 days to 36 months of age with suspected pneumococcal disease
MeSH Terms: interventions — Blood Culture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Bacterial isolates
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children with suspected pneumococcal invasive disease
  Interventions: Procedure: Blood culture; Procedure: Other cultures per Clinical routine practice

INTERVENTIONS:
Procedure: Blood culture — A baseline blood culture will be obtained in all participants
Procedure: Other cultures per Clinical routine practice — Cultures from other sterile sites will be obtained per routine clinical practice

SUMMARY:
Streptococcus pneumoniae is a major cause of pneumonia, sepsis, bacteremia and pneumococcal meningitis among infants and children worldwide. Knowledge of the epidemiology of pneumococcal disease is essential to assess the potential usefulness of pneumococcal disease usefulness of pneumococcal conjugate immunization. There is a paucity of information regarding pneumococcal disease burden in children in Latin America. Most studies are based on passive microbiology laboratory surveillance that does not capture all invasive disease, thus underestimating the true disease burden. Data from an active surveillance is available from an specific region in Costa Rica, before introduction of universal vaccination with PCV-7. On January 2009, PCV-7 was introduce into the universal vaccination program for all children born after or on September 2008 using a 3+1 regimen therefore there is a possibility to analyze the benefits of the introduction of this vaccine into the universal immunization program. The only effectiveness data from Latin America have been published from Uruguay where a significant decline in the incidence of pneumonias and meningitis was observed following the introduction of PCV-7. This was associated with an increment of serotypes 19A, 1,5 and 7F. Uruguay modify PCV-7 to PCV-13. In Costa Rica on August 2011, PCV-7 was changed for PCV 13. This study will provide information regarding the impact of PCV-7 and PCV-13.

DETAILED DESCRIPTION:
Study Objective(s):

Primary Objectives:

1. Determine the population-based incidence of invasive pneumococcal disease (IPD) defined as isolation of S. pneumoniae from a normally sterile site in children 28 days to 36 months of age with signs and symptoms of disease
2. Describe the serotype distribution of invasive S. pneumoniae isolates
3. Compare the incidence and serotype distribution of S. pneumoniae infection in the study population before and after universal introduction of the heptavalent conjugated vaccine against S. pneumoniae.

Secondary Objectives:

1. Describe the antibiotic resistance rates of invasive S. pneumoniae isolates
2. Describe the serotype distribution of resistant S. pneumoniae isolates
3. Assess the neurologic sequelae of pneumococcal meningitis
4. Describe the bacteriology other than S. pneumoniae

Study Design:

A prospective, population-based epidemiologic study in Costa Rica that will include children 28 days to 36 months of age presenting to or referred to a participant healthcare center with a temperature > or equal to 39.0 Celcius and/or clinical suspicion of pneumonia, meningitis, sepsis or other invasive pneumococcal disease regardless of temperature. Children who meet study entry criteria will be offered enrollment in the study. Informed consent will be obtained.

Data to be collected upon enrollment include: date of birth, race, sex, enrollment diagnosis, history of receipt of pneumococcal conjugate vaccine (PCV) and/or pneumococcal polysaccharide vaccine, residence, absence/presence of factors known to be associated with IPD: antibiotic use in the previous 7 days, daycare attendance, smokers in the household, > or equal 5 individuals in the household and presence of an underlying medical illness or chronic condition such: as sickle cell disease or other hemoglobinopathies, prematurity, HIV, immunodeficiency, reactive airways disease, systemic steroid use, neoplastic disease, pulmonary conditions, renal condition, cardiac condition, hematologic condition and/or diabetes.

One blood culture will be collected upon enrollment, before antibiotic administration if clinically possible. Specimens fro other sterile sites i.e, pleural fluid, CSF and joint fluid, will be collected as per routine medical practice. All bacteriology samples will undergo bacterial culture at the local laboratory for identification of pathogens, according to standard methodology. Bacterial isolates other than S. pneumoniae will be identify according to established standard microbiologic procedures. All other bacterial isolates will be store as per laboratory protocol for future microbiologic investigation. All S. pneumoniae isolates will be subcultured and sent on transport medium to a central laboratory for confirmation of identification, serotyping and antimicrobial susceptibility testing. Serotyping will be performed using type specific sera by Quellung reaction.

Results of cultures will be documented for all subjects. Final diagnosis and vital status will be collected on day 10 or hospital discharge, whichever occurs first, for all hospitalized subjects, all subjects whose culture (s) yield S. pneumoniae, and/or subjects whose inclusion criteria include clinical suspicion of meningitis.For subjects with suspected pneumonia, results of chest radiographs performed as part of normal standard of care taken 72 hours prior to or post study enrollment will be recorded as normal or abnormal and, if abnormal, presence of lobar consolidation, pleural effusion, both or other will be documented. The investigator will use World Health Organization (WHO) guidelines(Standardization of interpretation of chest radiographs for the diagnosis of pneumonia in children, from the World Health Organization Pneumonia Vaccine Trial Investigators'Group) to document the radiograph report on the subject's case report form. For subjects enrolled with suspected meningitis, final diagnosis will be documented. If meningitis is the final diagnosis it will be recorded as follows:

* Definite pneumococcal meningitis: Isolation of S. pneumoniae from the CSF, or from a blood culture of subject with >10 white blood cells (WBCs)/μL on examination of CSF and either CSF protein >100 mg/dL or CSF glucose <40 mg/dL or glucose CSF-to-serum ratio less than 0.6.
* Probable pneumococcal meningitis: CSF with >10 WBCs/μL and either other evidence suggestive of pneumococcal infection, such as Gram stain of CSF with gram-positive cocci or positive latex agglutination for S. pneumoniae in the CSF or any other non culture techniques; or isolation of S. pneumoniae in the blood of a subject admitted for suspected meningitis but lacking the CSF characteristics for definite pneumococcal meningitis, or CSF not obtained.
* Meningitis not pneumococcal: Evidence of meningitis (>10 WBCs/μL on examination of CSF and either CSF protein >100 mg/dL or CSF glucose < 40 mg/dL or glucose CSF-to-serum ratio less than 0.6) with isolation of another pathogen (not S. pneumoniae) from CSF or blood or with sterile cultures. For the subset of subjects identified with probable or definite pneumococcal meningitis, a neurologic examination will be conducted by a qualified physician for evaluation of neurologic sequelae between 6 and 9 months after enrollment to assess if the subject has any neurologic deficits secondary to their meningitis. Abnormalities may include, but are not limited to: vegetative state, mental retardation, brain damage, hydrocephalus, cerebral palsy, hearing impairment, vision impairment, seizures, and development delay. In participants subjects, if possible, a remnant of sterile fluids (example: CSF, joint, peritoneal, pleural fluid or other sterile fluid) will be collected and store at -70C for future testing designed only for identification of S. pneumoniae.

Duration of Study:

This study will be completed in approximately 09 months with the possibility of extending the trial for another year. Enrollment will last 09 months.

Number of Subjects:

Approximately 4000 children between the ages of 28 days and 36 months will be enrolled during the study period.

Diagnosis and Main Criteria for Inclusion:

1. Children 28 days to 36 months of age
2. Presenting to or referred to a participating healthcare facility with a measured temperature of ≥39.0 °C within 24 hours prior to screening, or with clinical suspicion of pneumonia, meningitis, sepsis, or other invasive pneumococcal disease, regardless of temperature
3. Subject belongs to the country specific target population for this study
4. Informed consent obtained from parent(s) or legal guardian(s)

Main Criteria for Exclusion:

1. Children younger than 28 days or older than 36 months of age at enrollment
2. Children suspected of having dengue fever as determined by local standard of care(i.e., platelet count, tourniquet test)

Safety Evaluation:

1. Subjects will be observed for 15 minutes after the blood culture is obtained for determination of protocol-related adverse effects.
2. Protocol-related adverse events and protocol related serious adverse events occurring within 1 day after blood collection will be reported based on local legislation on adverse event reporting.

Statistical Analysis:

The primary analysis will be the annual age-specific incidence rate of IPD estimated based on the number of identified cases from study sites and the size of the population at risk for children aged 28 days to 36 months in the same area. Ninety-five percent (95%) confidence intervals will be calculated based on the assumption of a Poisson distribution.

Descriptive analysis of serotype distributions for all IPD and individual S. pneumoniae infections, as well as for antimicrobial-resistant isolates will be performed. Summary data will be also be analyzed to assess the effects of age and other demographics as well as risk factors (described in-study-design) on IPD incidence and pneumococcal serotype distribution. Pooled analysis may be performed.

Rationale for Number of Subjects:

Based on published studies conducted in Latin America, the incidence of IPD in children less than 5 years of age varies widely (2.92/100,000 to 129/100,000). Based on the first ear analysis of protocol 0887XI-900 (april 20, 2007 - april 19, 2008) the documented incidence of IPD in the study area was 40.0 per 100,000 in children aged 28 days to less than 36 months with a peak incidence of 106.6/100,000 in children aged 28 days to less than 6 months of age. Furthermore, during the same period the incidence of chest radiograph confirmed pneumonia was 412.8 per 100,000 children aged 28 days to less than 36 months with a peak incidence of 744/100.000 children less than 12 months of age.

During that period the S. pneumoniae isolates obtained were: 14 (3), 6A (2) and one of the following: 3, 4, 6B, 7C, 9V 15B, 22F, 23 F. Because this study design represents a continuation of a similar study in the same area, with the only intervention been the universal application of the conjugated heptavalent vaccine to all newborns using a 3 + 1 regimen, we expect, after one year of universal vaccination, a decline of approximately 20% in the number of chest radiograph confirmed pneumonia, a 20% decline in the overall incidence of IPD and a 40% reduction in the incidence of IPD produced by vaccine type S.

pneumoniae isolates.

Ethical Considerations:

This study will be conducted in accordance with applicable Costa Rican law and regulations including, but not limited to, the International Conference on Harmonisation Guideline for Good Clinical Practice (GCP) and the ethical principles that have their origins in the Declaration of Helsinki. The institutional review board (IRB)/independent ethics committee (IEC) must review and approve the protocol and informed consent form (ICF) before any subjects are enrolled. The subject's parent(s) or legal guardian(s) must complete the informed consent process using the approved ICF before any procedures specified in the protocol are performed.

ELIGIBILITY:
Inclusion Criteria:

1. Children 28 days to 36 months of age
2. Presenting to or referred to a participating healthcare facility with a measured temperature of ≥39.0 °C within 24 hours prior to screening, or with clinical suspicion of pneumonia, meningitis, sepsis, or other invasive pneumococcal disease, regardless of temperature
3. Subject belongs to the country specific target population for this study
4. Informed consent obtained from parent(s) or legal guardian(s) -

Exclusion Criteria:

1. Children younger than 28 days or older than 36 months of age at enrollment
2. Children suspected of having dengue fever as determined by local standard of care(i.e., platelet count, tourniquet test) -

Ages: 28 Days to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Costa Rican children aged 28 days to 36 months of age with suspected pneumococcal invasive disease
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Impact of PCV 7 and PCV 13 on invasive pneumococcal disease in Costa Rican Children | 24 months

SECONDARY OUTCOMES:
Describe serotype distribution, antimicrobial susceptibility, neurological sequelae in children with meningitis and describe bacteriology other than S. pneumoniae | 30 months
Describe the antibiotic resistant rates of invasive S. pneumoniae isolates | 24 months
Describe the serotype distribution of resistant S. pneumoniae isolates | 24 months
Assess the neurologic sequelae of pneumococcal meningitis | 30 months
Describe the bacteriology other than S. pneumoniae | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Abdelnour, MD, Principal Investigator — Instituto de Atencion Pediatrica
Locations (5):
- Costa Rica (5):
  - Clinica Santa Catalina, Desamparados, Provincia de San José
  - Hospital CIMA San Jose, Escazú, Provincia de San José
  - Instituto de Atencion Pediatrica, San José, Provincia de San José
  - Hospital Clinica Biblica, San José, Provincia de San José
  - Hospital Metropolitano, San José, Provincia de San José